CLINICAL TRIAL: NCT04632524
Title: Evaluation of the Role of Low Dose Magnesium Sulfate in Anesthesia for Toxic Goiter Resection: A Randomized Controlled Trial
Brief Title: Evaluation of the Role of Low Dose Magnesium Sulfate in Anesthesia for Toxic Goiter Resection
Acronym: Anesthesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fayoum University Hospital (Other)
Responsible Party: Principal Investigator, Atef Mohamed Sayed mahmoud, Principal investigator, Fayoum University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: R68
Record Dates: First submitted 2020-08-30; First posted 2020-11-17 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Haemodynamic Stability
Keywords: Thyrotoxic goiter; heamodynamics; magnesium sulphate

STUDY DESIGN:
Intervention Model Description: sixty (60) patients ASA ǀ &ǁ patients of both sex aging 16-78 years (with primary or secondary thyrotoxic goiter and will be presented for thyroidectomy) will be allocated into one of two groups: Group (M) n=30 will receive Mg So4 pre-induction as an intravenous bolus 20mg/kg over 10 minutes and maintenance dose intraoperative 5/mg/kg/h intravenous and discontinued just before the end of the surgery. Group (S) n=30 will receive saline in equal volume.
Who Masked: Investigator
Masking Description: The patients were randomly allocated by a computer-generated table into one of two study groups. The randomization sequence was concealed in opaque sealed envelopes. The envelopes were opened by the study investigators just after recruitments and admission to the operation room.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MgSO4 (Active Comparator): Group (Mg So4) n=30 will receive Mg So4 pre-induction as an intravenous bolus 20mg/kg over 10 minutes and maintenance dose intraoperative 5/mg/kg/h intravenous and discontinued just before the end of the surgery.
  Interventions: Drug: MgSO4
- Placebo (Placebo Comparator): Group (P) n=30 will receive saline in equal volume. The surgeon , anesthesiologist and the person who will collect the data will be blinded for the prepared solution. The solution will be prepared by an expert anesthesia nurse
  Interventions: Drug: MgSO4

INTERVENTIONS:
Drug: MgSO4 — Group (M) n=30 will receive Mg So4 pre-induction as an intravenous bolus 20mg/kg over 10 minutes and maintenance dose intraoperative 5/mg/kg/h intravenous and discontinued just before the end of the surgery. Group (S) n=30 will receive saline in equal volume. The surgeon , anesthesiologist and the person who will collect the data will be blinded for the prepared solution. The solution will be prepared by an expert anesthesia nurse.

SUMMARY:
Anesthesia for toxic goiter removal is a challenging because of of hemodynamic instability especially during induction, intubation, manipulations of the gland, after removal of the gland and during emergence. So, hemodynamic stability is required all through the operation and even in the first 12 hours of the postoperative period to protect against complications e.g., hypertension, tachycardia, myocardial ischemia, bleeding and thyrotoxic crisis.Mg sulphate used in blunting pressor response during laryngoscopy and intubation. Also it was used in controlled hypotension technique. Also it was reported in decreasing postoperative nausea, vomiting, shivering and postoperative complications compared to controlled group.

DETAILED DESCRIPTION:
Patients and Methods:

After obtaining the approval of the Ethical Committee number (R68) of Al Fayoum University Hospitals and written informed consent from the patients, sixty (60) patients ASA ǀ &ǁ patients of both sex aging 20-70 years (with primary or secondary thyrotoxic goiter and will be presented for thyroidectomy) will be allocated into one of two groups: Group (M) n=30 will receive Mg So4 pre-induction as an intravenous bolus 20mg/kg over 10 minutes and maintenance dose intraoperative 5/mg/kg/h intravenous and discontinued just before the end of the surgery. Group (S) n=30 will receive saline in equal volume. The surgeon , anesthesiologist and the person who will collect the data will be blinded for the prepared solution. The solution will be prepared by an expert anesthesia nurse.

ELIGIBILITY:
Inclusion Criteria:

1. patients ASA ǀ &ǁ
2. patients of both sex
3. Aging from 20-70years
4. Pstients with primary or secondary thyrotoxic goiter

Exclusion Criteria:

1. Major hepatic disease
2. renal disease.
3. Cardiac dysfunction e.g. (heart Failure).
4. Uncontrolled hypertension
5. Advanced Ischemic heart diseases.
6. Known allergy to Mg So4.
7. Morbid obesity & pregnancy.
8. History of neuromuscular diseases.
9. cerebrovascular diseases.
10. Diabetic neuropathy.
11. patients receiving magnesium. supplementations.
12. Mental retardation
13. Patients on antiepileptic treatment
14. patients antipsychotics.
15. Hug goiter with retrosternal extension.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-10-16 (Actual); Primary Completion 2022-01-20 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
Blood pressure intraoperative | 5 minutes after induction of anesthesia
  Mean arterial blood pressure measurement in mmHg
Oxygen saturation intraoperative | 5 minutes after induction of anesthesia
  SPO2 Measurement as percentage (%)
Heart Rate intraoperative | 5 minutes after induction of anesthesia
  HR intraoperative beats per minutes
Blood pressure postoperative | 10minutes after extubation
  Mean arterial blood pressure measurement mmHg
Heart Rate postoperative | 10 minutes after extubation
  Heart Rate measurement by beats per minutes
Oxygen saturation postoperative | 10 minutes after extubation
  Spo2 measured as percentage %

SECONDARY OUTCOMES:
Sedation score post operative | 1 hour post operative
  Sedation score frome 0 point awake and alert to 4 non arousable
Visual analog scale postoperative(hrs) | 4 hours post operative
  A scale for measuring pain from 0 no pain up to 10 worst unbearable pain
Total opoid consumption intraoperative | 10 minutes after induction of anesthesia
  Total dose calculated
Serum Mg level at the beginning of operation | 10 minutes after induction of anesthesia
  Blood sample for measuring mg serum level
Total opoid consumption postoperative | 4 hours post operative
  Total dose calculated postoperative
Serum Mg level at the end of operation | 10 minutes befor extubation
  Blood sample for measuring mg serum level

CONTACTS AND LOCATIONS:
Locations (1):
- Atef, Al Fayyum, Egypt

IPD SHARING:
Plan to Share IPD: No
Email inquiry

REFERENCES:
- [Result] Alessandro Bacuzzi, Gianlorenzo Dionigi, Andrea Del Bosco, Giovanni Cantone, Tommaso Sansone, Erika Di Losa, Salvatore Cuffari. Anaesthesia for thyroid surgery: Perioperative management. International Journal of Surgery (2008);6: S82-S85. Sang-Hawn Do. Magnesium: a versatile drug for anesthesiologists. Korea J Anesthesiology 2013; 65 (1):4-8. Tramer MR, Shneider j, Marti RA, Rifat K. Role of magnesium sulfate in postoperative analgesia. Anesthesiology 1996; 84:340-7. Ryu JH, Sohn IS, Do SH. Controlled hypotension for middle ear surgery: a comparison between remifentanil and magnesium sulphate. Br J Anaesth 2009; 103: 490-5.